CLINICAL TRIAL: NCT05253027
Title: Foreign Body Swallows With Airway Affection in Pediatrics
Brief Title: Foreign Body Swallows in Pediatrics
Status: Completed | Type: Observational
Sponsor: Bahaa Mohammed Refaie (Other)
Responsible Party: Sponsor-Investigator, Bahaa Mohammed Refaie, lecturer of anesthesia and ICu, Sohag University
Organization: Sohag University (Other)
Other Study IDs: 2023
Record Dates: First submitted 2021-11-09; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Foreign Body in Oropharynx
Keywords: Foreign Bodies; Child; Respiratory distress; Hypopharynx; Esophagoscopy
MeSH Terms: conditions — Foreign Bodies; Dyspnea

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Foreign Body Ingestion (FBI) is a common clinical emergency in children. Most FBs smoothly pass through the digestive tract without complications; nevertheless, some FBs can cause severe morbidity and mortality. The current work aimed at evaluating how FBI can cause respiratory distress and stridor as well as their severity according to age, gender, lodgment site, and type of the object. Factors influencing morbidity and mortality among studied patients will be deliberated as well.

DETAILED DESCRIPTION:
Background: Foreign Body Ingestion (FBI) is a common clinical emergency in children. Most FBs smoothly pass through the digestive tract without complications; nevertheless, some FBs can cause severe morbidity and mortality. The current work aimed at evaluating how the FBI can cause respiratory distress and stridor as well as their severity according to age, gender, lodgment site, and type of the object. Factors influencing morbidity and mortality among studied patients will be deliberated as well.

Methods: It is a hospital-based descriptive study where all children between birth and 16 years of age who were admitted from January 1 st, 2018 to December, 31th 2021 for FBs removal were analyzed. All cases were subjected to complete history taking, physical, radiological, and bronchoscopic examination.

ELIGIBILITY:
Inclusion Criteria:

* children between birth and 16 years of age FBs removal
* history suggestive of foreign body swallow

Exclusion criteria:

- none

Ages: 1 Day to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children between birth and 16 years of age
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Respiratory distress | 24 hour after presentation
  stridor due to foreign body swallow

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided